CLINICAL TRIAL: NCT00855673
Title: Intermittent Mechanical Compression For Peripheral Arterial Disease
Acronym: FM-S1
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario Getafe (Other)
Responsible Party: Joaquin deHaro, Hospital Universitario Getafe
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FM-S1
Record Dates: First submitted 2009-03-02; First posted 2009-03-04 (Estimated); Last update posted 2009-03-04 (Estimated); Status verified 2009-02

CONDITIONS: Peripheral Arterial Disease
Keywords: Claudication; Peripheral Arterial Disease; Intermittent Compression; Mechanical Compression; Flowmedic
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental): Active group receiving intermittent compression
  Interventions: Device: Intermittent Mechanical Compression
- Control (Active Comparator): Standard Medical Treatment
  Interventions: Drug: Control

INTERVENTIONS:
Device: Intermittent Mechanical Compression — FM220 device
  Arms: Active
Drug: Control — Standard medical treatment
  Arms: Control

SUMMARY:
The study tests the use of a portable mechanical compression device (FM220, Flowmedic, USA) for the treatment of claudication and peripheral arterial disease.

Major endpoints are improved exercise tolerance and relevant blood pressure ratios

ELIGIBILITY:
Inclusion Criteria:

* stable claudication with an absolute claudication distance >40 meters but <300
* resting ABI in the affected limb <0.8

Exclusion Criteria:

* presence of diabetes

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2001-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
exercise tolerance | 3 months

SECONDARY OUTCOMES:
ankle-brachial index | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Joaquin DeHaro, MD, Principal Investigator — Hospital Universitario Getafe